CLINICAL TRIAL: NCT05040828
Title: Early Intervention With Leukotriene Receptor Antagonists in Patients With Grass Pollinosis: Effects on Clinical Symptoms and Allergic Inflammation
Brief Title: Early Intervention in Allergic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TR-Early intervention
Record Dates: First submitted 2021-08-25; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Allergic Rhinitis Due to Weed Pollen; Montelukast
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Early interventional treatment group (Experimental): The patients in this group:oral drug therapy from onset of the low pollen stage (August 1st, 2020) to the end of the pollen stage (September 30, 2020). Intranasal corticosteroids (mometasone furoate) from the high pollen stage (August 14, 2020) to the end of the pollen stage (September 30, 2020).
  Interventions: Behavioral: Start taking Montelukast Sodium Tablets 10mg quaque die orally two weeks before peak pollen count.
- Post-onset treatment group (Active Comparator): The patients in this group: oral drug therapy after the high pollen stage (August 14, 2020) to the end of the pollen stage (September 30, 2020.). Intranasal corticosteroids (mometasone furoate) from the high pollen stage (August 14, 2020) to the end of the pollen stage (September 30, 2020).
  Interventions: Behavioral: Montelukast Sodium Tablets 10mg quaque die orally was administered after peak pollen count.
- Control group (Active Comparator): The patients in this group:Intranasal corticosteroids (mometasone furoate) from the high pollen stage (August 14, 2020) to the end of the pollen stage (September 30, 2020).
  Interventions: Drug: No oral drug therapy throughout the pollen period

INTERVENTIONS:
Behavioral: Start taking Montelukast Sodium Tablets 10mg quaque die orally two weeks before peak pollen count. — Start taking Montelukast Sodium Tablets 10mg quaque die orally two weeks before peak pollen count.Intranasal corticosteroids (mometasone furoate) 100μg was used in the group after peak pollen count.
  Arms: Early interventional treatment group
Behavioral: Montelukast Sodium Tablets 10mg quaque die orally was administered after peak pollen count. — 10mg quaque die orally was administered after peak pollen count.Intranasal corticosteroids (mometasone furoate) 100μg was used in the group after peak pollen count.
  Arms: Post-onset treatment group
Drug: No oral drug therapy throughout the pollen period — Intranasal corticosteroids (mometasone furoate) 100μg was used in the group after peak pollen count.
  Arms: Control group

SUMMARY:
As many as 250 million people suffer from allergic rhinitis in China, which has a large population, early use of drugs may help better control the symptoms.This study aimed to investigate the effects of early interventional treatment with the leukotriene receptor antagonist (LTRA) montelukast on seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* patients showed distinct nasal symptoms (rhinorrhea, congestion, itching, and sneezing), and demonstrated sensitization to one of the grass pollen allergens (Artemisia, Chenopodium, and Humulus scandens) with an immunoglobulin (Ig) E ≥ 0.7 IU/mL, measured using the Pharmacia UniCAP system (Thermo Fisher Scientific China Co., Ltd., Shanghai, China).
* had not received any therapies for AR or antibiotics for at least 4 weeks before their outpatient clinic visit prior to the study
* all of the subjects in the study reside in Beijing.

Exclusion Criteria:

* Patients diagnosed with bronchial asthma, suffering from rhinitis outside the pollen season, chronic sinusitis, deviated nasal septum, using specific immunotherapy, or participating in another drug efficacy trial during the 4-week period preceding the study.
* pregnant women and minors

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
The change of subjective AR symptoms | baseline, visit 1: 2 weeks prior to the high weed pollen stage, visit 2: high weed pollen stage, visit 3: 2 weeks after the high weed pollen stage.
  Symptom change before and after treatment was estimated by Visual analogue scale(VAS) symptom score. The VAS symptom scores ranged from 0 (asymptomatic) to 10 (very severe). The questionnaire included nasal symptoms: nasal congestion, nasal discharge, sneezing, and rhinocnesmus; eye symptoms: lacrimation, eye itching, eye redness, swelling, and ophthalmodynia; airway symptoms: wheezing, chest constriction, cough, labored breathing.

SECONDARY OUTCOMES:
The change of objective examination: nasal function | baseline, visit 1: 2 weeks prior to the high weed pollen stage, visit 2: high weed pollen stage, visit 3: 2 weeks after the high weed pollen stage.
  Eccovision acoustic rhinometry was used to measure the nasal cavity volume (NCV) according to standardized recommendations. Measurements of nasal volume were made from the first 2 cm (V2), the first 4 cm (V4), from the first 6 cm (V6), from the segment between 0 and 5 cm (V0-5), and the segment between 0 and 7 cm (V0-7) of the nose. All measurements were performed three times by the same operator, and nasal volumes were calculated as the sum of both nostrils24. In the current study, the change in the nasal cavity volume was measured at 2-5 cm, as this seems to be an important variable for mucosal changes.24 Nasal airway resistance (NAR) was measured by anterior active rhinomanometry in a quiet room at temperature of 25°C and humidity of 70%. NAR was measured at 75 Pa point (R75T).
The change of cytokine expression | baseline, visit 1: 2 weeks prior to the high weed pollen stage, visit 2: high weed pollen stage, visit 3: 2 weeks after the high weed pollen stage.
  Quantitative real-time reverse transcription PCR (qRT-PCR) was used to analyze the mRNA expression levels of the cytokines interleukin-4, interleukin-5, interleukin-13, leukotriene C4, RANTES, tumor necrosis factor-α, thymic stromal lymphopoietin, and EOTAXIN in the nasal mucosa before and after treatment. The qRT-PCR data were processed using the 2-△△CT method.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Luo, Principal Investigator — Beijing Institute of Otolaryngology
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China